CLINICAL TRIAL: NCT07040891
Title: A Pilot Cluster Randomized Controlled Trial of "Just ASK™", an Intervention to Increase Discussions About Breast Cancer Clinical Trials
Brief Title: A Pilot Trial of "Just ASK™" to Increase Discussions About Breast Cancer Clinical Trials
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Carmen E. Guerra, Ruth C. and Raymond G. Perelman Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: BCRF-24-205
Record Dates: First submitted 2025-06-04; First posted 2025-06-27 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Just ASK training arm (Experimental): Participants in this arm will complete "Just ASK™" training, a web-based program designed to help providers understand the impact of assumptions about their patients' interest in cancer clinical trials and describe the "Just ASK™" framework for systematically asking all patients about cancer clinical trials.
  Interventions: Behavioral: Just ASK training
- Usual care arm (No Intervention): Participants in the usual care arm will not receive the training intervention.

INTERVENTIONS:
Behavioral: Just ASK training — "Just ASK™" is a web-based training designed to help providers understand the impact of assumptions about their patients' interest in cancer clinical trials. The training framework aims to increase clinical trial discussions with all cancer patients.
  Arms: Just ASK training arm

SUMMARY:
The goal of this study is to conduct a pilot cluster randomized controlled trial (RCT) of the "Just ASK™" training and implementation to increase provider discussion of cancer clinical trials (CCTs) with patients with breast cancer. The main research questions the study aims to answer are:

* Is a cluster RCT feasibility and acceptable? (This will inform the design of a future definitive cluster RCT)
* What are the determinants of the Just Ask training completion and implementation in practice to develop a better understanding for whom the intervention works, and under what circumstances?
* What are the discussion elements and approaches that are associated with participation in breast cancer clinical trials?

Researchers will compare the intervention arm (breast cancer clinics assigned to the Just ASK training) with the control arm (clinics receiving no training) to evaluate differences in clinical trial discussions with eligible breast cancer patients. Clinic participants in the intervention arm will complete the training and develop an implementation plan of training framework. Across all participating practices, up to 20 patient encounters per practice will be recorded to identify discussion elements associated with clinical trial participation.

ELIGIBILITY:
Inclusion criteria I (for oncology team members):

* Members of teams of oncology (physicians, nurses/nurse practitioners and coordinators) who routinely offer, consent and enroll patients in breast cancer clinical trials at the Abramson Cancer Center, Philadelphia, PA
* Able to provide informed consent.

Exclusion criteria I (for oncology team members):

- Previously completed "Just ASK™" training

Inclusion criteria II (for patient participants):

* Age >18
* New or relapsed patients diagnosed with breast cancer
* Are evaluated at the Abramson Cancer Center by those oncology team members participating in this study
* Are able to provide informed consent.

Exclusion criteria II (for patient participants):

- Already consented to participate in a breast cancer clinical trial for their treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Rates of discussion of breast cancer clinical trials | At the study completion (after all patient visit recordings are collected), an estimated average of 1 year after completion of recruitment.
  Will measure differences in rates of discussion of clinical trials with breast cancer patients between intervention and control arms

SECONDARY OUTCOMES:
Factors associated with breast cancer clinical trial participation (The outcome measure is qualitative in nature and does not involve quantitative variables. This will be a non-numeric outcome based on qualitative analysis of patient-provider encounters) | Up to 12 months after completion of data collection
  We will explore patient- and provider-level factors associated with breast cancer clinical trial participation. This will involve a qualitative analysis of audio-recorded patient visits from both study arms to identify recurring themes and contextual elements related to trial discussions. For example, factors such as geographic distance from the clinic or presence/absence of caregivers may influence a patient's decision to participate in clinical trials. However, we do not have a pre-defined set of measures for this qualitative study aim as the goal is to identify emergent themes through qualitative analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen E Guerra, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Castillo BS, Boehmer L, Schrag J, Howson A, Oyer R, Pierce L, Barrett NJ, Guerra CE. Oncologist-Reported Barriers and Facilitators to Offering Cancer Clinical Trials to Their Patients. Curr Oncol. 2024 May 28;31(6):3017-3029. doi: 10.3390/curroncol31060230. PMID 38920714
- [Background] Barrett NJ, Boehmer L, Schrag J, Benson AB 3rd, Green S, Hamroun-Yazid L, Howson A, Matin K, Oyer RA, Pierce L, Jeames SE, Winkfield K, Yang ES, Zwicker V, Bruinooge S, Hurley P, Williams JH, Guerra CE. An Assessment of the Feasibility and Utility of an ACCC-ASCO Implicit Bias Training Program to Enhance Racial and Ethnic Diversity in Cancer Clinical Trials. JCO Oncol Pract. 2023 Apr;19(4):e570-e580. doi: 10.1200/OP.22.00378. Epub 2023 Jan 11. PMID 36630671